CLINICAL TRIAL: NCT00685815
Title: Intravenous Iron Metabolism in Restless Legs Syndrome
Acronym: RLS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AG0117; 3P01AG021190 (NIH); 1VIT06013 (Other: American Regent)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2020-08

CONDITIONS: Restless Legs
Keywords: IV Iron; Restless Legs Syndrome; RLS; Iron
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric carboxymaltose (FCM) (Experimental): Intravenous iron (FCM)
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — 500mg FCM in 250cc normal saline (NS) IV over one hour, once on Day 3, once on Day 4
  Other Names: Injectafer
  Arms: Ferric carboxymaltose (FCM)
Drug: Placebo — 250cc normal saline (NS) IV over one hour, once on Day 3, once on Day 4
  Arms: Placebo

SUMMARY:
Double-blind, placebo-controlled, entitled: "Intravenous Iron Metabolism in Restless Legs Syndrome

DETAILED DESCRIPTION:
To determine the effects of high-dose infusions of iron on Restless Legs Syndrome (RLS) symptoms and brain concentrations of iron.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Restless Legs Syndrome (RLS).
* Presence of increased periodic leg movements of sleep (PLMS) before receiving treatment.
* Patient sleep times are between 9pm and 9am.
* Patient's RLS symptoms would occur daily if you were not on medication.

Exclusion Criteria:

* RLS secondary to other medical disorders as determined by history and physical/neurological examination.
* On a treatment (e.g., psychiatric medication) that might significantly alter RLS symptoms or study results and who cannot discontinue medication for the extended period of the study.
* History of multiple adverse drug reactions or specifically an allergy to IV iron.
* Currently experiencing a serious medical condition (chronic organ failure, active inflammation or infection, congestive heart failure, etc.) that might alter iron metabolism, would place them at risk, or interfere with study participation.
* An magnetic resonance imaging (MRI) is not possible because of medical reasons (Pacemaker; loose iron in the tissue) or concern about severe claustrophobia.
* Any condition that is likely to increase iron loss (chronic bleeding, excluding menstruation; medically necessary phlebotomy) or consumption (pregnancy).
* Serum ferritin >300mg/L or percent iron saturation >50%. This is to exclude subjects with probable hemochromatosis.
* Significant medical (e.g., inflammatory bowel syndrome; bowel dysmotility syndromes) or surgical (e.g., gastrojejunal bypass, colectomy) GI tract problems; and active chronic inflammatory processes (e.g., active hepatitis, rheumatoid arthritis, systemic lupus erythematosus). This is to exclude conditions which will potentially alter iron metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Earley, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Placebo: 250cc NS IV over one hour, once on Day 3, once on Day 4
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) | Placebo
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Groups:
- Ferric Carboxymaltose (FCM): Intravenous Iron (FCM)
  Ferric Carboxymaltose (FCM): 500mg FCM in 250cc NS IV over one hour, once on Day 3, once on Day 4
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) | Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Customized [Count of Participants; unit: Participants] — Age of Onset of RLS
  Participants
    < 25 years | 4 | 3 | 7
    25 - 50 years | 2 | 1 | 3
    > 50 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Duration Off Treatment
Description: Number of weeks that patients were able to remain off treatment for RLS
Time Frame: 2 weeks, 4 weeks, and 52 weeks
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Ferric Carboxymaltose (FCM) | Placebo
Number analyzed (Participants) | 8 | 4
participants
  Duration - 2 weeks | 6 | 3
  Duration - 20 weeks | 2 | 0
  Duration - 52 weeks | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: All events whether volunteered by the subject, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Ferric Carboxymaltose (FCM) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No